CLINICAL TRIAL: NCT06969586
Title: The Effect of Topical Rho-kinase (ROCK) Inhibitors on Corneas of Patients With Fuchs Endothelial Corneal Dystrophy (FECD)
Brief Title: The Effect of Topical Rho-kinase Inhibitors on Corneas of Patients With Fuchs Endothelial Corneal Dystrophy
Status: Enrolling by invitation | Type: Observational
Sponsor: University Hospital Dubrava (Other)
Responsible Party: Principal Investigator, Anđela Jukic, Principal Investigator, University Hospital Dubrava
Other Study IDs: 2025/0327-5
Record Dates: First submitted 2025-04-27; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Fuchs Endothelial Corneal Dystrophy; Cataract; Glaucoma
Keywords: Fuchs Endothelial Corneal Dystrophy (FECD); Rho-kinase inhibitors (ROCK); corneal edema; corneal endothelium
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy; Cataract; Glaucoma; Corneal Edema | interventions — netarsudil; Ophthalmic Solutions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- ROCK inhibitor group: Patients with Fuchs Endothelial Corneal Dystrophy and glaucoma scheduled for cataract surgery. ROCK inhibitor group will receive topical ROCK inhibitor for 30 days postoperatively.
  Interventions: Drug: Netarsudil 0.02% Ophthalmic Solution
- Placebo group: Patients with Fuchs Endothelial Corneal Dystrophy and glaucoma scheduled for cataract surgery. ROCK inhibitor group will receive topical placebo for 30 days postoperatively.
  Interventions: Drug: artificial tear substitute

INTERVENTIONS:
Drug: Netarsudil 0.02% Ophthalmic Solution — Topical Netarsudil 0.02% 1x daily for 30 days postoperatively
  Groups: ROCK inhibitor group
Drug: artificial tear substitute — Topical artificial tear substitute 1x daily for 30 days postoperatively.
  Groups: Placebo group

SUMMARY:
The goal of this study is to learn if topical ROCK inhibitors protect endothelial corneal cells in patients with glaucoma and Fuchs endothelial corneal dystrophy after cataract surgery. The main question it aims to answer is: do topical ROCK inhibitors decrease the loss of corneal endothelial cells after cataract surgery? Researchers will compare topical ROCK inhibitor to a placebo (a look-alike substance that contains no drug)

Participants will:

Take topical ROCK inhibitor or a placebo every day for 4 weeks after cataract surgery and visit the clinic for checkups and tests.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effect of topical Rho-kinase (ROCK) inhibitors on corneal endothelial cells (CECs) after cataract surgery in patients with cataract, glaucoma and Fuchs Endothelial Corneal Dystrophy (FECD). The study was approved by Ethics Committee of University Hospital Dubrava and will be conducted in accordance with tenets of the Declaration of Helsinki. Informed consent will be obtained from all individual participants included in the study.

Patients with glaucoma and FECD that require cataract surgery will be recruited. The inclusion criteria will be: age between 40 and 90 years; diagnosis of FECD and glaucoma; cataract grade II nuclear/cortical or posterior subcapsular (Lens Opacity Classification System III [LOCS III].

Exclusion criteria will be other anterior segment pathology (pseudoexfoliation syndrome, corneal opacities); ocular surface inflammation; intraoperative complications (posterior capsular rupture, vitreous loss, IOL not implanted in the capsular bag); previous ocular trauma or intraocular surgery.

Sample size was calculated to be 25 participants per group, using State statistical software (StataCorp LLC, College station, TX).

The patients will be randomized into two groups and the study drugs will be masked for both the patients and examiners. Group 1 will receive topical ROCK inhibitor netarsudil 0.02% ophthalmic solution 1x daily for four weeks after the surgery. Group 2 will receive topical placebo (artificial tear substitute) 1x daily for four weeks after the surgery. All patients will receive topical steroid antibiotic drops (dexamethasone, neomycin and polymyxin B, 1 mg, 3500 IU and 6000 IU/mL, respectively) four times daily for a week and then tapered over the next 3 weeks (three times daily for a week, then two times daily for a week and then one time daily for a week). All patients will be examined by a single researcher to limit observer bias. One experienced surgeon will performe all surgical procedures, which are consisted of topical anaesthesia, clear corneal small incision, capsulorhexis and phacoemulsification with the implantation of a foldable hydrophobic acrylic intraocular lens. At the end of the surgery, cefuroxime (1 mg) will be instilled into the anterior chamber. Phacoemulsification will be performed using CENTURION Vision System (Alcon Vision LLC, Fort Worth, TX). ECD (Endothelial Cell Density), CV (Coefficient of Variation) and % Hexagonal ( 6A or Hexagonality) will be determined using non contact specular microscope ( confocal endomicroscopy-530, Nidek Co, Ltd, Gamagori, Japan). Central corneal thickness (CCT) will be measured using ultrasound pachymetry (Micro Medical Devices, Inc, CA) and visual acuity will be evaluated using a Snellen chart and converted to logarithm of the minimum angle of resolution (LogMAR). Intraocular pressure (IOP) will be measured using Goldmann applanation tonometer (GAT). Measurements will be performed 7 days before the surgery and on 7th and 30th day postoperatively. Information on adverse effects will be collected for all patients during the study.

ELIGIBILITY:
Inclusion Criteria:

* age between 40 and 90 years;
* diagnosis of FECD and glaucoma;
* cataract grade II nuclear/cortical or posterior subcapsular (Lens Opacity Classification System III [LOCS III].

Exclusion criteria:

* other anterior segment pathology (pseudoexfoliation syndrome, corneal opacities);
* ocular surface inflammation;
* intraoperative complications (posterior capsular rupture, vitreous loss, IOL not implanted in the capsular bag);
* previous ocular trauma or intraocular surgery

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with glaucoma and FECD scheduled for cataract surgery.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Endothelial cell density (ECD) | 37 days
  ECD (Endothelial Cell Density) will be determined using non contact specular microscope ( confocal endomicroscopy-530, Nidek Co, Ltd, Gamagori, Japan).

SECONDARY OUTCOMES:
Visual acuity (VA) | 37 days
  Visual acuity (VA) will be measured using Snellen chart.

CONTACTS AND LOCATIONS:
Overall Officials: Josip Pavan, prof.dr.sc., Study Director — University Hospital Dubrava
Locations (1):
- University Hospital Dubrava, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No
There are no plans to share IPD due to privacy concerns and lack of participant consent for data sharing.